CLINICAL TRIAL: NCT06210750
Title: A Randomized Phase 2 Trial to Evaluate the Efficacy of BCL-2 Inhibitor Therapy With Chemotherapy Compared to Chemotherapy Alone in Adult Patients With Newly Diagnosed T-Cell ALL and T-Cell Lymphoblastic Lymphoma
Brief Title: Adding Targeted Drugs to Usual Chemotherapy for Adults With Newly Diagnosed T-Cell Acute Lymphoblastic Leukemia (T-ALL) and T-Cell Lymphoblastic Lymphoma (T-LBL)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Other - Protocol moved to Disapproved
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-09521; NCI-2023-09521 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2306 (Other: SWOG); S2306 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2024-01-17; First posted 2024-01-18 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: T Acute Lymphoblastic Leukemia; T Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Specimen Handling; Biopsy; calaspargase pegol; Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Spinal Puncture; Mercaptopurine; azathiopurine; Methotrexate; merphos; navitoclax; nelarabine; pegaspargase; Magnetic Resonance Spectroscopy; Thioguanine; venetoclax; Vincristine; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Arm 1 (AALL0434 regimen) (Active Comparator): See detailed description for Arm 1
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Procedure: Echocardiography; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Nelarabine; Drug: Pegaspargase; Procedure: Positron Emission Tomography; Drug: Thioguanine; Drug: Vincristine; Procedure: X-Ray Imaging
- Arm 2 (AALL0434 regimen with venetoclax) (Experimental): See detailed description for Arm 2
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Procedure: Echocardiography; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Nelarabine; Drug: Pegaspargase; Procedure: Positron Emission Tomography; Drug: Thioguanine; Drug: Venetoclax; Drug: Vincristine; Procedure: X-Ray Imaging
- Arm 3 (AALL0434 regimen with navitoclax) (Experimental): See detailed description for Arm 3
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Procedure: Echocardiography; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Biological: Navitoclax; Drug: Nelarabine; Drug: Pegaspargase; Procedure: Positron Emission Tomography; Drug: Thioguanine; Drug: Vincristine; Procedure: X-Ray Imaging
- Arm 4 (AALL0434 regimen with venetoclax and navitoclax) (Experimental): See detailed description for Arm 4
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Procedure: Echocardiography; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Biological: Navitoclax; Drug: Nelarabine; Drug: Pegaspargase; Procedure: Positron Emission Tomography; Drug: Thioguanine; Drug: Venetoclax; Drug: Vincristine; Procedure: X-Ray Imaging
- Arm 5 (AALL0434 [no nelarabine]) (Active Comparator): See detailed description for Arm 5
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Procedure: Echocardiography; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Pegaspargase; Procedure: Positron Emission Tomography; Drug: Thioguanine; Drug: Vincristine; Procedure: X-Ray Imaging
- Arm 6 (AALL0434 [no nelarabine] + navitoclax & venetoclax) (Experimental): See detailed description for Arm 6
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Procedure: Echocardiography; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Biological: Navitoclax; Drug: Nelarabine; Drug: Pegaspargase; Procedure: Positron Emission Tomography; Drug: Thioguanine; Drug: Venetoclax; Drug: Vincristine; Procedure: X-Ray Imaging
- Arm 7 (AALL0434 regimen) (Active Comparator): See detailed description for Arm 7
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Procedure: Echocardiography; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Nelarabine; Drug: Pegaspargase; Procedure: Positron Emission Tomography; Drug: Thioguanine; Drug: Vincristine
- Arm 8 (Remission induction with venetoclax and navitoclax) (Experimental): See detailed description for Arm 8
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Doxorubicin; Procedure: Echocardiography; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Biological: Navitoclax; Drug: Nelarabine; Drug: Pegaspargase; Procedure: Positron Emission Tomography; Drug: Thioguanine; Drug: Venetoclax; Drug: Vincristine; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Calaspargase Pegol — Given IV
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol-mknl; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
Drug: Cytarabine — Given IT, IV or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Navitoclax — Given PO
  Other Names: A-855071.0; ABT-263; BcI-2 Family Protein Inhibitor ABT-263
  Arms: Arm 3 (AALL0434 regimen with navitoclax); Arm 4 (AALL0434 regimen with venetoclax and navitoclax); Arm 6 (AALL0434 [no nelarabine] + navitoclax & venetoclax); Arm 8 (Remission induction with venetoclax and navitoclax)
Drug: Nelarabine — Given IV
  Other Names: 2-Amino-6-methoxypurine arabinoside; 506U78; Arranon; Compound 506U78; GW506U78
  Arms: Arm 1 (AALL0434 regimen); Arm 2 (AALL0434 regimen with venetoclax); Arm 3 (AALL0434 regimen with navitoclax); Arm 4 (AALL0434 regimen with venetoclax and navitoclax); Arm 6 (AALL0434 [no nelarabine] + navitoclax & venetoclax); Arm 7 (AALL0434 regimen); Arm 8 (Remission induction with venetoclax and navitoclax)
Drug: Pegaspargase — Given IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
  Arms: Arm 2 (AALL0434 regimen with venetoclax); Arm 4 (AALL0434 regimen with venetoclax and navitoclax); Arm 6 (AALL0434 [no nelarabine] + navitoclax & venetoclax); Arm 8 (Remission induction with venetoclax and navitoclax)
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
Procedure: X-Ray Imaging — Undergo X-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray
  Arms: Arm 1 (AALL0434 regimen); Arm 2 (AALL0434 regimen with venetoclax); Arm 3 (AALL0434 regimen with navitoclax); Arm 4 (AALL0434 regimen with venetoclax and navitoclax); Arm 5 (AALL0434 [no nelarabine]); Arm 6 (AALL0434 [no nelarabine] + navitoclax & venetoclax); Arm 8 (Remission induction with venetoclax and navitoclax)

SUMMARY:
This phase II trial tests the safety and effectiveness of giving chemotherapy with or without venetoclax and/or navitoclax for the treatment of patients with newly diagnosed T-cell acute lymphoblastic leukemia (T-ALL) or T-cell lymphoblastic lymphoma (T-LBL). Chemotherapy drugs work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax and navitoclax are in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. They may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving chemotherapy with or without venetoclax and/or navitoclax may be effective treatments for patients with newly diagnosed T-ALL or T-LBL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of venetoclax + navitoclax + AALL0434 chemotherapy backbone (arm 4) before initiating randomization. (Cohort 1) II. To compare rates of undetectable measurable residual disease (MRD) at day 29 following induction therapy of AALL0434 chemotherapy (arm 1) versus: 1) venetoclax + AALL0434 chemotherapy backbone (arm 2); 2) navitoclax + AALL0434 chemotherapy backbone (arm 3) and; 3) venetoclax and navitoclax + AALL0434 chemotherapy backbone (arm 4) (3 primary comparisons). (Cohort 1) III. To evaluate the safety of AALL0434 chemotherapy backbone (without nelarabine). (Cohort 2) IV. If the AALL0434 chemotherapy backbone is found to be safe, then to evaluate the safety of the backbone + venetoclax and navitoclax. (Cohort 2) V. To estimate the percent of participants with detectable disease in the bone marrow as measured by multiparameter flow cytometry at diagnosis. (Cohort 2) VI. To estimate rates of undetectable MRD at day 29 following induction therapy within and across treatment arms in cohort 2. (Cohort 2) VII. To evaluate the safety of modified AALL0434 chemotherapy backbone (including nelarabine). (Cohort 3) VIII. If the AALL0434 chemotherapy backbone is found to be safe, then to evaluate the safety of the backbone + venetoclax and navitoclax. (Cohort 3) IX. To estimate rates of undetectable MRD at day 29 within and across treatment arms in cohort 3. (Cohort 3)

SECONDARY OBJECTIVES:

I. To estimate the response rates of complete remission (CR), complete remission with incomplete count recovery (CRi), both with and without MRD, event-free survival, relapse-free survival, and overall survival across participant cohorts and within randomized regimens in cohort 1.

II. To estimate the frequency and severity of toxicities across participant cohorts and within randomized regimens in cohort 1.

III. Within cohorts 1-3, to evaluate the association of CR, CRi, event-free survival, relapse-free survival, and overall survival with the T-cell immunologic subtype of early T-cell precursor (ETP) lymphoblastic leukemia, defined as CD3+, CD7+, CD8-, CD1a-, and one or more myeloid/stem cell markers CD34, CD117, HLA-DR, CD13, CD33, CD11b, and CD65, but negative for myeloperoxidase (MPO).

IV. Within cohorts 1-3, to evaluate the association of endpoints (CR, CRi, event-free survival, relapse-free survival, and overall survival) with pretreatment characteristics (including age, gender, white blood cell count, central nervous system [CNS] leukemia at diagnosis, immunophenotype, karyotype).

V. Across cohorts 1-3 where laboratory data is available (laboratory evaluation is not mandated in the study), to evaluate serum asparaginase activity levels at day 8 and day 15 of Induction, at day 19 and day 26 of consolidation, and day 6 and 13 of interim maintenance courses, of reduced doses peg-asparaginase in participants age > 30 years and/or participants with at least one of the following risk factors for toxicity: body mass index (BMI) > 30, history of liver disease, history of diabetes mellitus type 2. To compare asparaginase activity levels between the different arms of cohort 1.

VI. Across cohorts 1-3, to estimate the frequency and severity of toxicities associated with reduced doses of peg-asparaginase in participants age > 30 years and/or in participants with at least one of risk factors for toxicity as noted above.

TRANSLATIONAL MEDICINE PRIMARY OBJECTIVE:

I. Across all cohorts, to estimate rates of MRD (day 29) with centrally evaluated flow cytometry.

TRANSLATIONAL MEDICINE SECONDARY OBJECTIVES:

I. Across all cohorts, to estimate rates of MRD (day 78 for cohorts 1 & 3, day 57 for cohort 2) with centrally evaluated flow cytometry.

II. Within and across cohorts 1-3, to estimate the percentage of participants with ETP and non-ETP immunophenotype.

III. Within and across cohorts 1-3, to evaluate the association of CR/CRi, event-free survival, relapse-free survival, and overall survival with ETP and non-ETP immunophenotype.

BANKING OBJECTIVE:

I. Across cohorts 1-3, to bank specimens for future correlative studies.

OUTLINE:

SAFETY PHASE: Patients in Cohort 1 are assigned to Arm 4. Patients in Cohort 2 are assigned to Arm 5 or Arm 6. Patients in Cohort 3 are assigned to Arm 7 or Arm 8.

RANDOMIZED PHASE: Patients in Cohort 1 are randomized to Arms 1, 2, 3, or 4.

ARM 1:

INDUCTION: Patients receive cytarabine intrathecally (IT) on day 1, vincristine intravenously (IV) and daunorubicin IV on days 1, 8, 15 and 22, dexamethasone orally (PO) twice per day (BID) on days 1-7 and 15-21, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on day 4, and methotrexate IT on days 8 and 29 (days 15 and 22 for patients with central nervous system [CNS 3] disease). Treatment continues for one 4-week cycle (weeks 1-4) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments.

CONSOLIDATION: Patients receive nelarabine IV on days 1-5 and 43- 47, cyclophosphamide IV on days 8 and 50, cytarabine IV or subcutaneously (SC) on days 8-11, 15-18, 50-53 and 57-60, mercaptopurine PO on days 8-21 and 50-63, vincristine IV on days 22, 29, 64, and 71, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 22 and 64 and methotrexate IT on days 15, 22, 57 and 64 (NOTE: Patients with CNS 3 disease omit methotrexate on day 22). Treatment continues for one 11-week cycle (weeks 6-16) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments. Patients who are MRD negative proceed, patients who are MRD positive are removed from the study.

INTERIM MAINTENANCE: Patients receive methotrexate IV and vincristine IV on days 1, 11, 21, 31 and 41, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 2 and 22 and methotrexate IT on days 1 and 31. Treatment continues for one 8-week cycle (weeks 17-24) in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION: Patients receive dexamethasone PO BID on days 1-7, and 15-21, doxorubicin IV on days 1, 8 and 15, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 4 and 50, nelarabine IV on days 29-33, cyclophosphamide IV on day 36, cytarabine IV or SC on days 36-39 and 43-46, thioguanine PO on days 36-49, vincristine IV on days 1, 8, 15, and 50 and methotrexate IT on days 1, 36, and 43. Treatment continues for one 9-week cycle (weeks 25-33) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive vincristine IV on days 1 and 57 of each cycle, dexamethasone PO BID on days 1-5, and 57-61 of each cycle, mercaptopurine PO on days 1-28 and 36-84 of each cycle, methotrexate PO on days 8, 15, 22, 36, 43, 50, 57, 64, 71, and 78 of each cycle, methotrexate IT on day 1 of each cycle, and nelarabine IV on days 29-33 of cycles 1-3. Cycles repeat every 84 days for a total of 2 years from the start of Interim Maintenance in the absence of disease progression or unacceptable toxicity.

Patients undergo x-ray and EKG at screening and echocardiogram or mitigated acquisition scan (MUGA), computed tomography (CT), positron emission tomography (PET), bone marrow aspiration, bone marrow biopsy, lumbar puncture and blood sample collection throughout the study.

ARM 2:

INDUCTION: Patients receive cytarabine IT on day 1, venetoclax PO on days 1-14, vincristine IV and daunorubicin IV on days 1,8,15 and 22, dexamethasone PO BID on days 1-7 and 15-21, peg-L-asparaginase IV on day 4 and methotrexate IT on days 8 and 29 (days 15 and 22 for patients with CNS 3 disease). Treatment continues for one 4-week cycle (weeks 1-4) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments.

CONSOLIDATION: Patients receive nelarabine IV on days 1-5 and 43 -47, cyclophosphamide IV on days 8 and 50, cytarabine IV on days 8-11, 15-18, 50-53 and 57-60, mercaptopurine PO on days 8-21 and 50-63, vincristine IV on days 22, 29, 64, and 71, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 22 and 64, methotrexate IT on days 15, 22, 57 and 64 (NOTE: Patients with CNS 3 disease omit methotrexate on day 22), and venetoclax PO on days 8-21. Treatment continues for one 11-week cycle (weeks 6-16) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments. Patients who are MRD negative proceed, patients who are MRD positive are removed from the study.

INTERIM MAINTENANCE: Patients receive methotrexate IV and vincristine IV on days 1, 11, 21, 31 and 41, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 2 and 22 and methotrexate IT on days 1 and 31. Treatment continues for one 8-week cycle (weeks 17-24) in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION: Patients receive dexamethasone PO BID on days 1-7, and 15-21, doxorubicin IV on days 1, 8 and 15, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 4 and 50, nelarabine IV on days 29-33, cyclophosphamide IV on day 36, cytarabine IV on days 36-39 and 43-46, thioguanine PO on days 36-49, vincristine IV on days 1, 8, 15, and 50 and methotrexate IT on days 1, 36, and 43. Treatment continues for one 9-week cycle (weeks 25-33) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive vincristine IV on days 1 and 57 of each cycle, dexamethasone PO BID on days 1-5, and 57-61 of each cycle, mercaptopurine PO on days 1-28 and 36-84, methotrexate PO on days 8, 15, 22, 36, 43, 50, 57, 64, 71, and 78 of each cycle, methotrexate IT on day 1 of each cycle, and nelarabine IV on days 29-33 of cycles 1-3. Cycles repeat every 12 weeks (84 days) for a total of 2 years from the start of Interim Maintenance in the absence of disease progression or unacceptable toxicity.

Patients undergo x-ray and EKG at screening and echocardiogram or MUGA, CT, PET, bone marrow aspiration, bone marrow biopsy, lumbar puncture and blood sample collection throughout the study.

ARM 3:

INDUCTION: Patients receive cytarabine IT on day 1, vincristine IV and daunorubicin IV on days 1, 8, 15 and 22, dexamethasone PO BID on days 1-7 and 15-21, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on day 4, navitoclax PO on days 1-14 and methotrexate IT on day 8 and 29 (days 15 and 22 for patients with CNS 3 disease). Treatment continues for one 4-week cycle (weeks 1-4) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments.

CONSOLIDATION: Patients receive nelarabine IV on days 1-5 and 43 -47, cyclophosphamide IV on days 8 and 50, cytarabine IV on days 8-11, 15-18, 50-53 and 57-60, mercaptopurine PO on days 8-21 and 50-63, vincristine IV on days 22, 29, 64, and 71, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 22 and 64, navitoclax PO on days 8-21 and methotrexate IT on days 15, 22, 57 and 64 (NOTE: Patients with CNS 3 disease omit methotrexate on day 22). Treatment continues for one 11-week cycle (weeks 6-16) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments. Patients who are MRD negative proceed, patients who are MRD positive are removed from the study.

INTERIM MAINTENANCE: Patients receive methotrexate IV and vincristine IV on days 1, 11, 21, 31 and 41, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 2 and 22 and methotrexate IT on days 1 and 31. Treatment continues for one 8-week cycle (weeks 17-24) in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION: Patients receive dexamethasone PO BID on days 1-7, and 15-21, doxorubicin IV on days 1, 8 and 15, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 4 and 50, nelarabine IV on days 29-33, cyclophosphamide IV on day 36, cytarabine IV on days 36-39 and 43-46, thioguanine PO on days 36-49, vincristine IV on days 1, 8, 15, and 50 and methotrexate IT on days 1, 36, and 43. Treatment continues for one 9-week cycle (weeks 25-33) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive vincristine IV on days 1 and 57 of each cycle, dexamethasone PO BID on days 1-5, and 57-61 of each cycle, mercaptopurine PO on days 1-28 and 36-84 of each cycle, methotrexate PO on days 8, 15, 22, 36, 43, 50, 57, 64, 71, and 78 of each cycle, methotrexate IT on day 1 of each cycle, and nelarabine IV on days 29-33 of cycles 1-3. Cycles repeat every 12 weeks (84 days) for a total of 2 years from the start of Interim Maintenance in the absence of disease progression or unacceptable toxicity.

Patients undergo x-ray and EKG at screening and echocardiogram or MUGA, CT, PET, bone marrow aspiration, bone marrow biopsy, lumbar puncture and blood sample collection throughout the study.

ARM 4:

INDUCTION: Patients receive cytarabine IT on day 1, vincristine IV and daunorubicin IV on days 1, 8, 15 and 22, dexamethasone PO BID on days 1-7 and 15-21, peg-L-asparaginase and calaspargase pegol-MKNL IV on day 4, venetoclax PO and navitoclax PO on days 1-14 and methotrexate IT on day 8 and 29 (days 15 and 22 for patients with CNS 3 disease). Treatment continues for one 4-week cycle (weeks 1-4) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments.

CONSOLIDATION: Patients receive nelarabine IV on days 1-5 and 43 -47, cyclophosphamide IV on days 8 and 50, cytarabine IV on days 8-11, 15-18, 50-53 and 57-60, mercaptopurine PO on days 8-21 and 50-63, vincristine IV on days 22, 29, 64, and 71, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 22 and 64, navitoclax PO and venetoclax PO on days 8-21 and methotrexate IT on days 15, 22, 57 and 64 (NOTE: Patients with CNS 3 disease omit methotrexate on day 22). Treatment continues for one 11-week cycle (weeks 6-16) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments. Patients who are MRD negative proceed, patients who are MRD positive are removed from the study.

INTERIM MAINTENANCE: Patients receive methotrexate IV and vincristine IV on days 1, 11, 21, 31 and 41, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 2 and 22 and methotrexate IT on days 1 and 31. Treatment continues for one 8-week cycle (weeks 17-24) in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION: Patients receive dexamethasone PO BID on days 1-7, and 15-21, doxorubicin IV on days 1, 8 and 15, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 4 and 50, nelarabine IV on days 29-33, cyclophosphamide IV on day 36, cytarabine IV on days 36-39 and 43-46, thioguanine PO on days 36-49, vincristine IV on days 1, 8, 15, and 50 and methotrexate IT on days 1, 36, and 43. Treatment continues for one 9-week cycle (weeks 25-33) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive vincristine IV on days 1 and 57 of each cycle, dexamethasone PO BID on days 1-5, and 57-61 of each cycle, mercaptopurine PO on days 1-28 and 36-84 of each cycle, methotrexate PO on days 8, 15, 22, 36, 43, 50, 57, 64, 71, and 78 of each cycle, methotrexate IT on day 1 of each cycle, and nelarabine IV on days 29-33 of cycles 1-3. Cycles repeat every 12 weeks (84 days) for a total of 2 years from the start of Interim Maintenance in the absence of disease progression or unacceptable toxicity.

Patients undergo x-ray and EKG at screening and echocardiogram or MUGA, CT, PET, bone marrow aspiration, bone marrow biopsy, lumbar puncture and blood sample collection throughout the study.

ARM 5:

INDUCTION: Patients receive cytarabine IT on day 1, vincristine IV and daunorubicin IV on days 1, 8, 15 and 22, dexamethasone PO BID on days 1-7 and 15-21, peg-L-asparaginase and calaspargase pegol-MKNL IV on day 4 and methotrexate IT on day 8 and 29 (days 15 and 22 for patients with CNS 3 disease). Treatment continues for one 4-week cycle (weeks 1-4) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments.

CONSOLIDATION: Patients receive cyclophosphamide IV on days 1 and 29, cytarabine IV or SC on days 1-4, 8-11, 29-33, and 36-39, mercaptopurine PO on days 1-14 and 29-42, vincristine IV on days 15, 22, 43, and 50, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 15 and 43, and methotrexate IT on days 1, 8, 15 and 22 (NOTE: Patients with CNS 3 disease omit methotrexate on days 15 and 22). Treatment continues for one 8-week cycle (weeks 6-13) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments. Patients who are MRD negative proceed, patients who are MRD positive are removed from the study.

INTERIM MAINTENANCE: Patients receive methotrexate IV and vincristine IV on days 1, 11, 21, 31 and 41, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 2 and 22 and methotrexate IT on days 1 and 31. Treatment continues for one 8-week cycle (weeks 14-21) in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION: Patients receive dexamethasone PO BID on days 1-7and 15-21, doxorubicin IV on days 1, 8 and 15, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 4 and 43, cyclophosphamide IV on day 29, cytarabine IV or SC on days 29-32 and 36-39, thioguanine PO on days 29-42, vincristine IV on days 1, 8, 15, 43 and 50, and methotrexate IT on days 1, 29, and 36. Treatment continues for one 9-week cycle (weeks 22-30) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive vincristine IV on days 1, 29 and 57 of each cycle, dexamethasone PO BID on days 1-5, 29-33, and 57-61 of each cycle, mercaptopurine PO on days 1-84 of each cycle, methotrexate PO on days 8, 15, 22, 36, 43, 50, 57, 64, 71, and 78 of each cycle, and methotrexate IT on day 1 of each cycle. Cycles repeat every 12 weeks (84 days) for a total of 2 years from the start of Interim Maintenance in the absence of disease progression or unacceptable toxicity.

Patients undergo x-ray and EKG at screening and echocardiogram or MUGA, CT, PET, bone marrow aspiration, bone marrow biopsy, lumbar puncture and blood sample collection throughout the study.

ARM 6:

INDUCTION: Patients receive cytarabine IT on day 1, vincristine IV and daunorubicin IV on days 1, 8, 15 and 22, dexamethasone PO BID on days 1-7 and 15-21, peg-L-asparaginase and calaspargase pegol-MKNL IV on day 4, venetoclax PO and navitoclax PO on days 1-14 and methotrexate IT on day 8 and 29 (days 15 and 22 for patients with CNS 3 disease). Treatment continues for one 4-week cycle (weeks 1-4) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments.

CONSOLIDATION: Patients receive cyclophosphamide IV on days 1 and 29, cytarabine IV on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO on days 1-14 and 29-42, vincristine IV on days 15, 22, 43 and 50, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 15 and 43, navitoclax PO and venetoclax PO on days 1-14 and methotrexate IT on days 1, 8, 15 and 22. Treatment continues for one 8-week cycle (weeks 6-13) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments. Patients who are MRD negative proceed, patients who are MRD positive are removed from the study.

INTERIM MAINTENANCE: Patients receive methotrexate IV and vincristine IV on days 1, 11, 21, 31 and 41, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 2 and 22 and methotrexate IT on days 1 and 31. Treatment continues for one 8-week cycle (weeks 14-21) in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION: Patients receive dexamethasone PO BID on days 1-7, and 15-21, doxorubicin IV on days 1, 8 and 15, peg-L-asparaginase IV and calaspargase pegol-MKNL IV on days 4 and 43, cyclophosphamide IV on day 29, cytarabine IV on days 29-32, and 36-39, thioguanine PO on days 29-42, vincristine IV on days 1, 8, 15, 43 and 50 and methotrexate IT on days 1, 29, and 36. Treatment continues for one 9-week cycle (weeks 22-30) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive vincristine IV on days 1, 29 and 57 of each cycle, dexamethasone PO BID on days 1-5, 29-33, and 57-61 of each cycle, mercaptopurine PO on days 1-84 of each cycle, methotrexate PO on days 8, 15, 22, 36, 43, 50, 57, 64, 71, and 78 of each cycle, and methotrexate IT on day 1 of each cycle. Cycles repeat every 12 weeks (84 days) for a total of 2 years from the start of Interim Maintenance in the absence of disease progression or unacceptable toxicity.

Patients undergo x-ray and EKG at screening and echocardiogram or MUGA, CT, PET, bone marrow aspiration, bone marrow biopsy, lumbar puncture and blood sample collection throughout the study.

ARM 7:

INDUCTION: Patients receive cytarabine IT on day 1, vincristine IV and daunorubicin IV on days 1, 8, 15 and 22, dexamethasone PO BID on days 1-7, peg-L-asparaginase IV on day 15, and methotrexate IT on day 8 and 29 (days 15 and 22 for patients with CNS 3 disease). Treatment continues for one 4-week cycle (weeks 1-4) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments.

CONSOLIDATION: Patients receive nelarabine IV on days 1-5 and 43-47, cyclophosphamide IV on days 8 and 50, cytarabine IV or SC on days 8-11, 15-18, 50-53, and 57-60, mercaptopurine PO on days 8-21, and 50-63, vincristine IV on days 22, 29, 64, and 71, peg-L-asparaginase IV on days 22 and 64, and methotrexate IT on days 15, 22, 57 and 64 (NOTE: Patients with CNS 3 disease omit methotrexate on day 22). Treatment continues for one 11-week cycle (weeks 6-16) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments. Patients who are MRD negative proceed, patients who are MRD positive are removed from the study.

INTERIM MAINTENANCE: Patients receive methotrexate IV and vincristine IV on days 1, 11, 21, 31 and 41, peg-L-asparaginase IV on days 2 and 22 and methotrexate IT on days 1 and 31. Treatment continues for one 8-week cycle (weeks 17-24) in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION: Patients receive dexamethasone PO BID on days 1-7, doxorubicin IV on days 1, 8 and 15, peg-L-asparaginase IV, on days 4 and 50, nelarabine IV on days 29-33, cyclophosphamide IV on day 36, cytarabine IV or SC on days 36-39, and 43-46, thioguanine PO on days 36-49, vincristine IV on days 1, 8, 15, and 50 and methotrexate IT on days 1, 36, and 43. Treatment continues for one 9-week cycle (weeks 25-33) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive vincristine IV on days 1 and 57 of each cycle, dexamethasone PO BID on days 1-5, and 57-61 of each cycle, mercaptopurine PO on days 1-28 and 36-84 of each cycle, methotrexate PO on days 8, 15, 22, 36, 43, 50, 57, 64, 71, and 78 of each cycle, methotrexate IT on day 1 of each cycle, and nelarabine IV on days 29-33 of cycles 1-3. Cycles repeat every 12-weeks (84 days) for a total of 2 years from the start of Interim Maintenance in the absence of disease progression or unacceptable toxicity.

Patients undergo x-ray and EKG at screening and echocardiogram or MUGA, CT, PET, bone marrow aspiration, bone marrow biopsy, lumbar puncture and blood sample collection throughout the study.

ARM 8:

INDUCTION: Patients receive cytarabine IT on day 1, vincristine IV and daunorubicin IV on days 1, 8, 15 and 22, dexamethasone PO BID on days 1-7, peg-L-asparaginase on day 15, venetoclax PO and navitoclax PO in days 1-14, and methotrexate IT on day 8 and 29 (days 15 and 22 for patients with CNS 3 disease). Treatment continues for one 4-week cycle (weeks 1-4) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments.

CONSOLIDATION: Patients receive nelarabine IV on days 1-5 and 43-47, cyclophosphamide IV on days 8 and 50, cytarabine IV on days 8-11, 15-18, 50-53, and 57-60, mercaptopurine PO on days 8-21, and 50-63, vincristine IV on days 22, 29, 64, and 71, peg-L-asparaginase IV on days 22 and 64, venetoclax PO and navitoclax PO on days 8-21, and methotrexate IT on days 15, 22, 57 and 64 (NOTE: Patients with CNS 3 disease omit methotrexate on day 22). Treatment continues for one 11-week cycle (weeks 6-16) in the absence of disease progression or unacceptable toxicity. Patients then undergo disease assessments. Patients who are MRD negative proceed, patients who are MRD positive are removed from the study.

INTERIM MAINTENANCE: Patients receive methotrexate IV and vincristine IV on days 1, 11, 21, 31 and 41, peg-L-asparaginase IV on days 2 and 22 and methotrexate IT on days 1 and 31. Treatment continues for one 8-week cycle (weeks 17-24) in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION: Patients receive dexamethasone PO BID on days 1-7, doxorubicin IV on days 1, 8 and 15, peg-L-asparaginase IV, on days 4 and 50, nelarabine IV on days 29-33, cyclophosphamide IV on day 36, cytarabine IV or SC on days 36-39, and 43-46, thioguanine PO on days 36-49, vincristine IV on days 1, 8, 15, and 50 and methotrexate IT on days 1, 36, and 43. Treatment continues for one 9-week cycle (weeks 25-33) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive vincristine IV on days 1 and 57 of each cycle, dexamethasone PO BID on days 1-5, and 57-61 of each cycle, mercaptopurine PO on days 1-28 and 36-84 of each cycle, methotrexate PO on days 8, 15, 22, 36, 43, 50, 57, 64, 71, and 78 of each cycle, methotrexate IT on day 1 of each cycle, and nelarabine IV on days 29-33 of cycles 1-3. Cycles repeat every 84 days for a total of 2 years from the start of interim maintenance in the absence of disease progression or unacceptable toxicity.

Patients undergo x-ray and EKG at screening and echocardiogram or MUGA, CT, PET, bone marrow aspiration, bone marrow biopsy, lumbar puncture and blood sample collection throughout the study.

After completion of study treatment, patients are followed up periodically for up to 10 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have newly diagnosed T-cell acute lymphoblastic leukemia (T-ALL) or T-lineage lymphoblastic lymphoma (T-LBL) based on 2022 World Health Organization (WHO) criteria. Participants with acute leukemia of ambiguous lineage (ALAL), including mixed phenotype acute leukemia (MPAL), are not eligible for this trial
* For T-ALL, immunophenotyping of the blood or marrow lymphoblasts must be performed by flow cytometry to confirm T-cell lineage and exclude ALAL or MPAL. Appropriate lineage-specific antigens include cytoplasmic or surface CD3 for T lineage, myeloperoxidase (MPO) or monocytic antigens (CD11c, CD14, CD64, lysozyme) for myeloid lineage, and CD19, CD20, CD22, CD79a, CD10 and PAX5 for B lineage. For T-LBL, immunohistochemistry on paraffin embedded tissue alone can be used to establish the diagnosis, although flow cytometry is preferred
* NOTE: Systemic chemotherapy must begin within 72 hours of first dose of intrathecal therapy
* Collection of pretreatment blood and bone marrow specimens must be completed within 14 days prior to registration for all participants. If bone marrow is unable to be aspirated and blood blast percentage is at least 5%, additional blood should be collected as instructed in the study calendar
* Participants must not have received prior induction chemotherapy for T-ALL/LBL. Prior treatments with hydroxyurea, all-trans retinoic acid (ATRA), corticosteroids, leukapheresis to reduce peripheral blast count and prevent complications from leukocytosis, and a single dose of intrathecal cytarabine and/or methotrexate with or without steroids are permitted
* Participants must discontinue strong CYP3A4 inducers within 7 days prior to registration. Dose adjustments for CYP3A4 inhibitors/inducers during protocol therapy are defined in the protocol
* Participants must be 18-60 years old
* Participants must have Zubrod/Eastern Cooperative Oncology Group (ECOG performance status of 0-2
* Participants must have a complete medical history and physical exam within 28 days prior to registration
* Participants with extramedullary disease at diagnosis must have a CT scan with contrast of chest, neck, abdomen, pelvis, or whole body to obtain baseline values within 28 days prior to registration
* Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN). Participants with history of Gilbert's disease or leukemia involving the liver must have total bilirubin ≤ 5 x institutional ULN within 7 days prior to registration
* Aspartate aminotransferase (AST)/ Alanine aminotransferase (ALT) Both must be ≤ 3 × institutional ULN unless related to leukemia involving the liver
* Participants must have a serum creatinine 1.5 ≤ the ULN OR measured OR calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault Formula. This specimen must have been drawn and processed within 7 days prior to registration
* Participants must have a lumbar puncture to determine CNS involvement of ALL within 14 days prior to registration. Intrathecal cytarabine and/or methotrexate administered prior to study registration may count as the first dose of intrathecal therapy required as part of protocol therapy
* Participants must have cardiac ejection fraction >= 50% by MUGA or 2-D echocardiogram within 28 days before registration. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to registration, if indicated
* Participants with known human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at registration and have undetectable viral load test on the most recent test results obtained within 6 months prior to registration
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to registration, if indicated
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial (in the opinion of the treating physician)
* Participants must not be pregnant or nursing. Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 24 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants with T-ALL must not have a history of seizure disorder due to nelarabine administration
* Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System
* Participants must agree to have blood and bone marrow specimens submitted for MRD

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-09 (Estimated); Primary Completion 2026-09-22 (Estimated); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (Cohorts 1, 2 and 3) | Up to 10 years
  National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events will be used to determine severity of toxicity.
Undetectable minimal residual disease (MRD) (Cohort 1) | At day 29 following induction
  There will be three primary analyses, each comparing an experimental arm with the shared control arm using Fisher's exact test with a one-sided alpha of 10%. All eligible randomized participants will be used in the efficacy comparison.
Percent of participants with detectable disease in the bone marrow (Cohort 2) | At diagnosis and at days 29 and 57
  Binomial estimates will be reported along with exact 95% confidence intervals.
Undetectable MRD (Cohorts 1 and 3) | At days 29 and 78
  Binomial estimates will be reported along with exact 95% confidence intervals.

SECONDARY OUTCOMES:
Rate of complete remission (CR) | End of consolidation therapy
  Response rates in each arm and cohort will be calculated and presented with exact binomial 95% confidence intervals.
Rate of complete remission with incomplete count recovery (CRi) with and without MRD | End of consolidation therapy
  Response rates in each arm and cohort will be calculated and presented with exact binomial 95% confidence intervals.
Event free survival | From the date of initial registration on study until the first of the following events: death from any cause, relapse from MRD-negative remission, or completion of protocol therapy without documentation of MRD-negative remission, up to 10 years
  Will be estimated using the method of Kaplan-Meier; randomized arms within Cohort 1 will be compared using the stratified log rank test.
Relapse free survival | From the date the participant first achieves CR or CRi until relapse from CR/CRi or death from any cause, up to 10 years
  Will be estimated using the method of Kaplan-Meier; randomized arms within Cohort 1 will be compared using the stratified log rank test.
Overall survival | From the day of registration to death from any cause, up to 10 years
  Will be estimated using the method of Kaplan-Meier; randomized arms within Cohort 1 will be compared using the stratified log rank test.
Incidence of adverse events | Up to 10 years
  National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events will be used to determine severity of toxicity.
Serum asparaginase activity levels | At day 8 and day 15 of induction, day 19 and 26 of consolidation and day 6 and 13 of interim maintenance
  Of patients with reduced doses Peg-asparaginase in participants age > 30 years and/or participants with at least one of the following risk factors for toxicity: Body mass index (BMI) > 30, history of liver disease, history of diabetes mellitus type 2.
Incidence of adverse events associated with reduced doses of Peg-asparaginase | Up to 10 years
  Participants age >30 years and/or in participants with at least one of risk factors for toxicity.

OTHER OUTCOMES:
Rates of MRD | At day 29 (all cohorts), day 78 (cohorts 1 and 3), and day 57 (cohort 2)
  With centrally evaluated flow cytometry. Binomial estimates will be reported along with exact 95% confidence intervals.
Percentage of participants with ETP and non-ETP immunophenotype | Diagnosis
  Binomial estimates will be reported along with exact 95% confidence intervals.
Association of CR/CRi, event-free survival, relapse-free survival, and overall survival with early thymic precursor (ETP) and non-ETP immunophenotype | Up to 10 years
  Response rates will be compared using Fisher's exact test.
  Survival outcomes will be compared using log-rank tests.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M O'Dwyer, Principal Investigator — SWOG Cancer Research Network

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm